CLINICAL TRIAL: NCT06790017
Title: Temperature Measurement for Transurethral Prostatectomy Surgery in Elderly Patient
Brief Title: Hemoglobin-to-red Blood Cell Distribution Width Ratio and Hypothermia for Elderly Patient
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Gokcen Kulturoglu, doctor, Ankara Etlik City Hospital
Other Study IDs: AESH-EK1-2024-0082
Record Dates: First submitted 2025-01-09; First posted 2025-01-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Transurethral Resection of Prostate Syndrome; Elderly (People Aged 65 or More); General Anesthetic
Keywords: elderly; hypothermia
MeSH Terms: conditions — Hypothermia | interventions — Body Temperature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low hemoglobin to red cell distribution width ratio (HRR): Patients whose HRR rate is below 9.97 and are considered frail
  Interventions: Other: body temperature
- High hemoglobin to red cell distribution width ratio (HRR): Patients whose HRR ratio is above 9.97 and are considered non-frail
  Interventions: Other: body temperature

INTERVENTIONS:
Other: body temperature — Body temperature measurement will be performed in the preoperative and intraoperative periods.

SUMMARY:
As individuals age, they often enter a phase of increased "frailty." Elderly and frail patients represent a population that requires heightened sensitivity and close monitoring during surgical procedures. This study aims to investigate the relationship between the Hemoglobin-to-Red Blood Cell Distribution Width (Hb/RDW) ratio and perioperative hypothermia in elderly patients undergoing transurethral prostatectomy. This is an observational study. Preoperative blood test results and intraoperative body temperature measurements of the patients will be recorded in our data forms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provided informed consent.
* Patients scheduled for transurethral prostatectomy surgery.
* Patients classified as ASA-PS 1, 2, or 3.
* Male patients aged 65 years or older.
* Patients undergoing elective surgery.
* Patients receiving general anesthesia.

Exclusion Criteria:

* Patients who did not provide informed consent.
* Patients undergoing emergency surgery.
* Patients with conditions that disrupt thermoregulation (e.g., intracranial mass, peripheral vascular diseases, sepsis).
* Patients with a body temperature of <34℃ or >38℃ upon arrival at the preoperative waiting room.
* Patients who used heating methods other than the routine cotton cover in the preoperative waiting room.
* Patients who received additional heating methods other than the routinely applied intraoperative hot air blower drapes.
* Patients undergoing surgery under any type of anesthesia other than general anesthesia.
* Patients who were taken out of the operating room while intubated.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Etlik City Hospital, Urology Operating Rooms
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Perioperative Hypothermia | 1 hour before anesthesia and intraoperative
  Perioperative hypothermia is defined as any core temperature less than 96.8°F (36.0°C)

SECONDARY OUTCOMES:
Frailty | preoperative
  The relationship between hemoglobin to red cell distribution width ratio (HRR) and frailty
Red blood cell distribution width | 1 hour before anesthesia and intraoperative
  The relationship between red blood cell distribution width (RDW) and hypothermia

CONTACTS AND LOCATIONS:
Overall Officials: Gokcen KULTUROGLU, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author, (GK). The data are not publicly available due to our participants' informed consent forms.

REFERENCES:
- [Background] Zhu M, Wei C, Yang X, Huang Y, Xu Y, Xiong Z. Lower haemoglobin-to-red blood cell distribution width ratio is independently associated with frailty in community-dwelling older adults: a cross-sectional study. BMJ Open. 2023 Jul 9;13(7):e069141. doi: 10.1136/bmjopen-2022-069141. PMID 37423632
- [Background] Qu J, Zhou T, Xue M, Sun H, Shen Y, Chen Y, Tang L, Qian L, You J, Yang R, Liu Y. Correlation Analysis of Hemoglobin-to-Red Blood Cell Distribution Width Ratio and Frailty in Elderly Patients With Coronary Heart Disease. Front Cardiovasc Med. 2021 Aug 27;8:728800. doi: 10.3389/fcvm.2021.728800. eCollection 2021. PMID 34513961